CLINICAL TRIAL: NCT01406223
Title: Mechanistic Evaluations of Pre-Cessation Therapies for Smoking Cessation
Acronym: ConNicBrain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00028331; 1P50DA027840-01A1 (NIH)
Record Dates: First submitted 2011-06-12; First posted 2011-08-01 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; Smoking cessation; Zyban; Chantix; Nicotine patches; varenicline; bupropion; fMRI
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation | interventions — Varenicline; Bupropion; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- varenicline (Active Comparator): For the first 3 days after being switched from Nicotine Replacement Therapy (NRT) occurring at one week before the target quit date, smokers in this group will receive varenicline at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week. Subsequently, the dose will be 1 mg twice per day, and will remain at that dose for the remainder of the 12 weeks. During the time they receive varenicline, smokers in this group will also receive placebo bupropion and placebo patches.
  Interventions: Drug: Varenicline; Drug: Nicotine patches; Other: Placebo bupropion; Other: Placebo patch
- NRT (nicotine patches only) (Active Comparator): 21 mg/24 h for 2 weeks before the quit date and 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. After the 1st week, smokers in this group will also receive placebo bupropion and placebo varenicline.
  Interventions: Drug: Nicotine patches; Other: Placebo varenicline; Other: Placebo bupropion
- varenicline + bupropion (Active Comparator): For the first 3 days after being switched from Nicotine Replacement Therapy (NRT) occurring at one week before the target quit date, smokers in this group will receive varenicline at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week plus bupropion at a dose of 150mg once per day. Subsequently, the dose of varenicline will be 1 mg twice per day and the dose of bupropion will be 150 mg twice per day, and will remain at that dose for the remainder of the 12 weeks. During the time they receive varenicline and bupropion, smokers in this group will also receive placebo patches.
  Interventions: Drug: Varenicline; Drug: Bupropion; Drug: Nicotine patches; Other: Placebo patch
- Post-quit NRT (Placebo Comparator): Nicotine patches at 21 mg/24 h for 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. After the 1st week, smokers in this group will also receive placebo bupropion and placebo varenicline.
  Interventions: Drug: Nicotine patches; Other: Placebo varenicline; Other: Placebo bupropion; Other: Placebo patch

INTERVENTIONS:
Drug: Varenicline
  Other Names: Chantix
  Arms: varenicline; varenicline + bupropion
Drug: Bupropion
  Other Names: Zyban
  Arms: varenicline + bupropion
Drug: Nicotine patches
  Other Names: Nicoderm
Other: Placebo varenicline
  Arms: NRT (nicotine patches only); Post-quit NRT
Other: Placebo bupropion
  Arms: NRT (nicotine patches only); Post-quit NRT; varenicline
Other: Placebo patch
  Arms: Post-quit NRT; varenicline; varenicline + bupropion

SUMMARY:
The purpose of this study is to look at brain function in order to understand how different treatments work to help people quit smoking. In this study, the investigators will look at the effects of nicotine patches, Chantix alone or Chantix paired with Zyban.

ELIGIBILITY:
Inclusion Criteria:

* Are generally healthy;
* Are 18-50 years old;
* Smoke an average of at least 10 cigarettes per day for at least three cumulative years;
* Have an afternoon expired air carbon monoxide (CO) reading of at least 10ppm;
* Are right-handed as measured by a two-item scale used in our laboratory;
* Express a desire to quit smoking in the next thirty days.
* Potential subjects must agree to use acceptable contraception during their participation in this study.

Potential subjects must agree to avoid the following during their participation in this study:

* participation in any other nicotine-related modification strategy outside of this protocol;
* use of tobacco products other than cigarettes, including pipe tobacco, cigars, e-cigarettes, snuff, and chewing tobacco;
* use of experimental (investigational) drugs or devices;
* use of illegal drugs;
* use of opiate medications.

Exclusion Criteria:

* Inability to attend all required experimental sessions;
* Presence of conditions that would make MRI unsafe (e.g. pacemaker);
* Hypertension (systolic >140 mm Hg, diastolic >100 mm Hg, coupled with a history of hypertension); subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100.
* Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg).
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pains (unless history, exam, and ECG clearly indicate a non-cardiac source);
* Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* History of skin allergy;
* Active skin disorder (e.g., psoriasis) within the last five years, except minor skin conditions (including but not limited to facial acne, minor localized infections, and superficial minor wounds);
* Liver or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Lung disorder (including but not limited to Chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes;
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Current psychiatric disease (with the exception of anxiety disorders, Obsessive-compulsive disorder (OCD) and Attention deficit hyperactivity disorder (ADHD));
* Bulimia or anorexia;
* Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
* Current depression;
* Pregnant or nursing mothers;
* Alcohol abuse;
* Significant adverse reaction to nicotine patch, bupropion/Wellbutrin/Zyban or Chantix/Varenicline in the past.
* Use (within the past 30 days) of:

  * Illegal drugs (or if the urine drug screen is positive);
  * Experimental (investigational) drugs;
  * Psychiatric medications including antidepressants, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
  * Smokeless tobacco (chewing tobacco, snuff), cigars or pipes;
  * Nicotine replacement therapy or any other smoking cessation aid.
* Use (within the past 14 days) of:

  * Opiate medications for pain or sleep (non-opiate medication for pain or sleep will be allowed).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 282 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Joseph McClernon, Ph.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Center for Nicotine and Smoking Cessation Research, Durham, North Carolina
  - Duke Center for Nicotine and Smoking Cessation Research, Raleigh, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 282 participants who were consented and screened, 191 were screen fails, 2 withdrew voluntarily before being assigned to a study arm, and 13 were lost to contact between screening and the first study visit. Therefore, only 76 participants were randomized and started the study.
Groups:
- Varenicline: For the first 3 days after being switched from Nicotine Replacement Therapy (NRT) occurring at one week before the target quit date, smokers in this group will receive varenicline at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week. Subsequently, the dose will be 1 mg twice per day, and will remain at that dose for the remainder of the 12 weeks. During the time they receive varenicline, smokers in this group will also receive placebo bupropion and placebo patches.
  Varenicline
  Nicotine patches
  Placebo bupropion
  Placebo patch
- NRT (Nicotine Patches Only): 21 mg/24 h for 2 weeks before the quit date and 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. After the 1st week, smokers in this group will also receive placebo bupropion and placebo varenicline.
  Nicotine patches
  Placebo varenicline
  Placebo bupropion
- Varenicline + Bupropion: For the first 3 days after being switched from Nicotine Replacement Therapy (NRT) occurring at one week before the target quit date, smokers in this group will receive varenicline at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week plus bupropion at a dose of 150mg once per day. Subsequently, the dose of varenicline will be 1 mg twice per day and the dose of bupropion will be 150 mg twice per day, and will remain at that dose for the remainder of the 12 weeks. During the time they receive varenicline and bupropion, smokers in this group will also receive placebo patches.
  Varenicline
  Bupropion
  Nicotine patches
  Placebo patch
- Post-quit NRT: Nicotine patches at 21 mg/24 h for 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. After the 1st week, smokers in this group will also receive placebo bupropion and placebo varenicline.
  Nicotine patches
  Placebo varenicline
  Placebo bupropion
  Placebo patch
Period: Overall Study
Arm/Group | Varenicline | NRT (Nicotine Patches Only) | Varenicline + Bupropion | Post-quit NRT
Started | 18 | 19 | 20 | 19
Completed | 6 | 7 | 2 | 3
Not Completed | 12 | 12 | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | NRT (Nicotine Patches Only) | Varenicline + Bupropion | Post-quit NRT | Total
Number analyzed (Participants) | 18 | 19 | 20 | 19 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 20 | 19 | 75
  >=65 years | 0 | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.56 (10.68) | 41.89 (12.22) | 38.35 (11.42) | 37.16 (10.59) | 38.75 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 8 | 10 | 40
  Male | 7 | 8 | 12 | 9 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 0 | 5
  Not Hispanic or Latino | 16 | 18 | 18 | 19 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 6 | 9 | 7 | 34
  White | 5 | 11 | 10 | 12 | 38
  More than one race | 1 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 20 | 19 | 76

OUTCOME MEASURES:

1. Primary Outcome: The Amygdala, Anterior Insula, and Medial Prefrontal Cortex Scans Will be Compared to Evaluate Significant Differences
Description: Mean blood-oxygen-level dependent (BOLD) contrast sensitive functional magnetic resonance imaging (fMRI) cue-reactivity signal following 2 week pre-quit treatment, controlling for baseline cue-reactivity.
Time Frame: change from baseline in whole brain blood-oxygen-level dependent (BOLD) contrast sensitive functional magnetic resonance imaging (fMRI) images collected during a cue-reactivity task following 2 weeks of pre-quit treatment
Population: Only participants who completed both scanning sessions and provided useable data were included in imaging analysis.
Measure: Mean (Standard Deviation); unit: percent BOLD signal change
Arm/Group | Varenicline | NRT (Nicotine Patches Only) | Varenicline + Bupropion | Post-quit NRT
Number analyzed (Participants) | 10 | 13 | 8 | 8
percent BOLD signal change
  left amygdala | 0.057 (0.285) | .007 (.186) | .160 (.258) | .129 (.278)
  right amydala | .051 (.337) | -.014 (.190) | .134 (.266) | .020 (.249)
  left anterior insula | .094 (.196) | .013 (.244) | -.015 (.160) | .179 (.288)
  right anterior insula | -.008 (.224) | .065 (.305) | .019 (.188) | .082 (.333)
  left medial prefrontal cortex | .129 (.162) | .026 (.294) | -.120 (.562) | .009 (.200)
  right medial prefrtonal cortex | .058 (.171) | -.010 (.277) | -.176 (.641) | -.017 (.178)

2. Secondary Outcome: Days to First Cigarette Following Quitting Smoking
Description: Days to first cigarette (i.e. lapse) will be measured via self-report.
Time Frame: Up to 11 weeks post quit day.
Population: Twenty-eight subjects dropped from the study prior to their scheduled quit day, so they were not included in these analyses.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Varenicline | NRT (Nicotine Patches Only) | Varenicline + Bupropion | Post-quit NRT
Number analyzed (Participants) | 13 | 14 | 10 | 11
days | 9.15 (22.143) | 15.21 (26.066) | 9.90 (23.960) | 5.73 (18.666)

ADVERSE EVENTS:
Time Frame: Subjects were receiving study drugs for 13 weeks.
Description: At each study session during this period subjects completed a questionnaire about side effects. Subjects were also told to contact us between study sessions if side effects were bothersome.
Arm/Group | Varenicline | NRT (Nicotine Patches Only) | Varenicline + Bupropion | Post-quit NRT
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 3/18 | 6/19 | 6/20 | 4/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=18) | NRT (Nicotine Patches Only) (N=19) | Varenicline + Bupropion (N=20) | Post-quit NRT (N=19)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Excessive Sweating (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 2 (7) | 1 (1) | 2 (3)
Thirst (General disorders) | 0 (0) | 2 (7) | 0 (0) | 3 (5)
Hiccups (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 3 (3) | 1 (2)
Joint/Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (7)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Irritability (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Nightmares (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vivid Dreams (Nervous system disorders) | 2 (3) | 1 (1) | 3 (6) | 3 (6)
Insomnia (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 3 (9)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Libido (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Itching/Burning at Patch Site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash at Patch Site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Mouth/Throat Irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upset Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Statistical comparisons of imaging data between groups are limited due to small sample size in each condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No